CLINICAL TRIAL: NCT03200951
Title: The Effect of Epidural Analgesia on Intracranial Pressure by Measuring the Optic Nerve Sheath Diameter Using Ultrasound in Pediatric Patients With Cerebral Palsy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 4-2017-0341
Record Dates: First submitted 2017-06-22; First posted 2017-06-27 (Actual); Last update posted 2018-10-29 (Actual); Status verified 2018-10

CONDITIONS: Cerebral Palsy
MeSH Terms: conditions — Cerebral Palsy | interventions — Anesthesia, Epidural

STUDY DESIGN:
Intervention Model Description: Randomly selected patients of the bolus group are given 0.3 ml/kg bolus of 0.15% ripivacaine for epidudral block. In contrast, patients in the infusion group are given 0.3 ml/kg/hr 0.15% ripivacaine for epidural block.
Who Masked: Participant, Investigator
Masking Description: Participants and investigator are blinded to group assignment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Bolus group (Experimental)
  Interventions: Drug: Bolus group for epidural block
- Infusion group (Active Comparator)
  Interventions: Drug: Infusion group for epidural block

INTERVENTIONS:
Drug: Bolus group for epidural block — Randomly selected patients of the bolus group are given 0.3 ml/kg bolus of 0.15% ripivacaine for epidural block.
  Other Names: ripivacaine
  Arms: Bolus group
Drug: Infusion group for epidural block — Randomly selected patients of the infusion group are given 0.3 ml/kg/hr 0.15% ripivacaine for epidural block.
  Other Names: ripivacaine
  Arms: Infusion group

SUMMARY:
Ultrasonography of optic nerve sheath diameter shows a good level of diagnostic accuracy for detecting intracranial hypertension. The aim of this study is to evaluate the effect of epidural block on intracranial pressure in pediatric patients with cerebral palsy undergoing osteotomy of lower extremity. Forty patients, aged 4 years to 13 years, receiving epidural block before osteotomy will be divided into bolus group (n=20) and infusion group (n=20). Randomly selected patients of the bolus group are given 0.3 ml/kg bolus of 0.15% ripivacaine for epidural block. In contrast, patients in the infusion group are given 0.3 ml/kg/hr 0.15% ripivacaine for epidural block. The primary endpoint is the difference in the optic nerve sheath diameter after epidural block measured by optic nerve ultrasonography between groups.

ELIGIBILITY:
Inclusion Criteria:

* Pediatric patients with cerebral palsy from 4 to 13 years of age undergoing osteotomy
* Body weight ≤ 40 kg

Exclusion Criteria:

* Patients with contraindications to epidural analgesia (local infection, clotting disorders, anatomical abnormalities, sepsis, etc.)
* Patients with symptoms or signs associated with a history of elevated intracranial pressure or elevated intracranial pressure
* Patients with ophthalmic disease or surgery
* The estimated operation time is less than 70 minutes.
* All parents of the subject are foreigners or illiterate

Ages: 4 Years to 13 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 40 (Actual)
Dates: Start 2017-08-22 (Actual); Primary Completion 2018-05-31 (Actual); Study Completion 2018-05-31 (Actual)

PRIMARY OUTCOMES:
The difference in the optic nerve sheath diameter(ONSD) between groups | 5 minutes before epidural block
  The optic nerve sheath diameter measured by optic nerve ultrasonography.
The difference in the optic nerve sheath diameter(ONSD) between groups | 1 second after epidural block
  The optic nerve sheath diameter measured by optic nerve ultrasonography.
The difference in the optic nerve sheath diameter(ONSD) between groups | 10 minutes after epidural block
  The optic nerve sheath diameter measured by optic nerve ultrasonography.
The difference in the optic nerve sheath diameter(ONSD) between groups | 70 minutes after epidural block
  The optic nerve sheath diameter measured by optic nerve ultrasonography.

SECONDARY OUTCOMES:
The difference in the number of patients whose ONSD values increased to more than 5.75 mm at each time point between the two groups | 5 minutes before epidural block
  The optic nerve sheath diameter measured by optic nerve ultrasonography
The difference in the number of patients whose ONSD values increased to more than 5.75 mm at each time point between the two groups | 1 second after epidural block
  The optic nerve sheath diameter measured by optic nerve ultrasonography
The difference in the number of patients whose ONSD values increased to more than 5.75 mm at each time point between the two groups | 10 minutes after epidural block
  The optic nerve sheath diameter measured by optic nerve ultrasonography
The difference in the number of patients whose ONSD values increased to more than 5.75 mm at each time point between the two groups | 70 minutes after epidural block
  The optic nerve sheath diameter measured by optic nerve ultrasonography

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Anesthesiology and Pain Medicine, Anesthesia and Pain Research Institue, Yonsei Universiy College of Medicine, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Lin Y, Li Q, Liu J, Yang R, Liu J. Comparison of continuous epidural infusion and programmed intermittent epidural bolus in labor analgesia. Ther Clin Risk Manag. 2016 Jul 14;12:1107-12. doi: 10.2147/TCRM.S106021. eCollection 2016. PMID 27471390
- [Background] Padayachy LC, Padayachy V, Galal U, Pollock T, Fieggen AG. The relationship between transorbital ultrasound measurement of the optic nerve sheath diameter (ONSD) and invasively measured ICP in children. : Part II: age-related ONSD cut-off values and patency of the anterior fontanelle. Childs Nerv Syst. 2016 Oct;32(10):1779-85. doi: 10.1007/s00381-016-3068-4. Epub 2016 Sep 20. PMID 27659820